CLINICAL TRIAL: NCT02948647
Title: Diets Based on PNPLA3 Genotype for Reducing Liver Fat in Hispanics With Pediatric Non-alcoholic Fatty Liver Disease
Brief Title: Healthy Eating Through Reduction Of Excess Sugar
Acronym: HEROES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-11-00446
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: NAFLD
Keywords: obesity; fatty liver; sugar; PNPLA3
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Fatty Liver | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Will receive standard of care, which is general dietary advice
- Intervention Group (Experimental): Will receive standard of care as well as sugar-reduction education
  Interventions: Other: Standard of care plus sugar-reduction education

INTERVENTIONS:
Other: Standard of care plus sugar-reduction education — This is a 12-week intervention where subjects will be educated on how to monitor their added sugar consumption. They will be asked to eliminate consumption of sweetened beverages for the 12-week period and will be receiving a weekly delivery of water bottles to their homes to displace the sweetened beverages in their home environment.
  Arms: Intervention Group

SUMMARY:
The purpose of the study is to determine the effect of dietary sugar reduction in obese children and examine whether there are differential effects based on genotype of a single amino acid substitution in the PNPLA3 gene that is highly prevalent in Hispanics and associated with significantly elevated liver fat.

DETAILED DESCRIPTION:
This dietary intervention aims at developing a more personalized and targeted treatment for NAFLD in Hispanic children and adolescents who are GG for the PNPLA3 variant. The investigators previous publications have shown that this particular demographic has a greater than 2-fold higher liver fat compared to GC and CC individuals. They have also demonstrated a significant gene*dietary sugar interaction with a significant association between liver fat and dietary sugar intake in GG subjects with no such association in GC or CC individuals. These studies suggests that different dietary strategies may have differential effects on reducing liver fat, depending on PNPLA3 genotype. To confirm this, the investigators will complete a clinical trial in 120 overweight and obese Hispanic children (12 - 18 years) with clinically verified NAFLD who will be randomized to one of two 12-week interventions:

Group 1 (standard of care control group): Dietary intervention focused on healthy eating (n=60; 30GG + 30GC/CC)

Group 2 (standard of care + sugar reduction): Dietary intervention based on healthy eating and sugar reduction focused on reduction of sugary beverages and added sugar towards a goal of 10% of daily calories (n=60; 30GG + 30GC/CC)

The following outcomes will be measured before and after intervention: Total liver fat fraction, and visceral and subcutaneous abdominal adipose tissue volume by magnetic resonance imaging (MRI); liver fibrosis by magnetic resonance elastography (MRE); total body fat by DEXA; liver enzymes, fasting insulin, glucose, lipids, free fatty acids and inflammatory markers, gut microbiome, and insulin and glucose response to an oral glucose challenge. The investigators hypothesize that liver fat fraction, liver fibrosis, and metabolic outcomes, such as fasting and 2h-glucose and insulin, and inflammatory biomarkers, will show significantly greater improvements with sugar reduction relative to control. In addition, the investigators also hypothesize a treatment*genotype interaction whereby the reduction in liver fat will be significantly greater in GG relative to CC/CG subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: This study is limited to Hispanics because of their higher risk of NAFLD, higher frequency (~50%) of the at-risk PNPLA3 allele (G), and because no prior studies have targeted improvement in liver fat and NAFLD in this high-risk population. As with all of our ongoing studies, Hispanic ethnicity will be based on self-identity for the participants as well as their parents and grandparents.
* Gender: Males and females will be eligible for this study.
* Age: Children 12 to 18 years of age will be eligible. In our experience, children younger than around 10 years of age and greater than 18 years would require different intervention/counseling strategies. Therefore, we can develop a more consistent "age-neutral" approach if we limit the age range to 12-18 years.
* Weight status: Subjects will be eligible if they are obese, defined by a BMI > 95th percentile for age and gender.

Exclusion Criteria:

* Diabetes: Presence of type 1 or 2 diabetes, as defined by fasting plasma glucose > 126 mg/dl, or positive for diabetes related antibodies including ICA512 and GAD. Participants testing positive for diabetes will be referred for treatment. Subjects with pre-diabetes will be eligible for the study
* Pregnancy: Women who self-report as pregnant or obtain a positive pregnancy test result during Visit 1 will be excluded. Furthermore, should a woman become pregnant during the course of the intervention, she will be withdrawn from the study at that time and asked to no longer participate. This is in order to protect the mother and child from radiation involved with the DEXA scan and potential complications associated with a low-sugar diet.
* Medication: Taking any medications known to influence liver function, insulin action or lipid levels
* Self-prescribed dietary supplements: Taking any non-prescription supplements that could potentially affect liver function and liver fat (eg vitamin E or fish oils)
* Other metabolic diseases: Diagnosis of other syndromes or diseases that may influence insulin action and secretion (e.g., maturity-onset diabetes of the young, lipoatrophic diabetes, cystic fibrosis), or body composition and fat distribution (e.g. Cushing syndrome, Down syndrome, lipodystrophy)
* Other medical condition: Previously diagnosed with any major illness since birth (e.g. severe intrauterine growth retardation, chronic birth asphyxia, cancer)
* Familial hyperlipidemia: Patients with a family history of hyperlipidemia will be excluded, due to the particular genetic background of this disease, which may bias our results. Familial hyperlipidemia will be defined as LDL/cholesterol > 160 mg/dL and/or triglycerides > 200 mg/dL in both the participant AND at least one family member (first degree: parents or siblings).
* Smoking or drinking: Self-reported current smoking participants (more than 1 cigarette in the past week) will be excluded due to the potential effect of smoking on weight control and inflammatory status. Consumption of alcohol on a regular basis (40g/day alcohol per day determined by questionnaire) will also be excluded due to its important role in liver disease. Use of recreational drugs will also be an exclusion criteria, due to the potent effect of cannabinoids receptors on weight status and food intake.
* Participation in a weight-loss or exercise program: participants who have participated to a weight-loss or exercise program in the past three months will be excluded due to its potential effect on weight status.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Total liver fat fraction by Magnetic resonance imaging (MRI) at baseline | Baseline
  Abdominal fat distribution (visceral fat versus subcutaneous abdominal fat), and liver fat fraction will be assessed by magnetic resonance imaging at the USC Radiology imaging center on a research-dedicated GE 3 Tesla scanner. Visceral adipose tissue, subcutaneous abdominal adipose tissue and fat in the entire liver will be determined using the 3D IDEAL method.
Total liver fat fraction by Magnetic resonance imaging (MRI) at 12 weeks | 12 weeks
  Abdominal fat distribution (visceral fat versus subcutaneous abdominal fat), and liver fat fraction will be assessed by magnetic resonance imaging at the USC Radiology imaging center on a research-dedicated GE 3 Tesla scanner. Visceral adipose tissue, subcutaneous abdominal adipose tissue and fat in the entire liver will be determined using the 3D IDEAL method.
Change in total liver fat fraction by Magnetic resonance imaging (MRI) from baseline to 12 weeks | Baseline and 12 weeks
  Abdominal fat distribution (visceral fat versus subcutaneous abdominal fat), and liver fat fraction will be assessed by magnetic resonance imaging at the USC Radiology imaging center on a research-dedicated GE 3 Tesla scanner. Visceral adipose tissue, subcutaneous abdominal adipose tissue and fat in the entire liver will be determined using the 3D IDEAL method.

SECONDARY OUTCOMES:
Liver fibrosis by Magnetic Resonance Enterography (MRE) at baseline | Baseline
  MRE is a non-invasive technology for measuring tissue stiffness that has been validated against liver fibrosis by biopsy; as liver stiffness by MRE increases systematically with fibrosis stage. MRE can also discriminate between patients with moderate and severe fibrosis (grades 2-4) and those with mild fibrosis (sensitivity, 86%; specificity, 85%). MRE will be performed during the same scan for adipose tissue on the research-dedicated 3.0 Tesla GE Scanner equipped with the Mayo Clinic MRE apparatus, and synchronized motion-encoded GRE sequence, based on published validation studies.
Liver fibrosis by Magnetic Resonance Enterography (MRE) at 12 weeks | 12 weeks
  MRE is a non-invasive technology for measuring tissue stiffness that has been validated against liver fibrosis by biopsy; as liver stiffness by MRE increases systematically with fibrosis stage. MRE can also discriminate between patients with moderate and severe fibrosis (grades 2-4) and those with mild fibrosis (sensitivity, 86%; specificity, 85%). MRE will be performed during the same scan for adipose tissue on the research-dedicated 3.0 Tesla GE Scanner equipped with the Mayo Clinic MRE apparatus, and synchronized motion-encoded GRE sequence, based on published validation studies.
Change in Liver fibrosis by Magnetic Resonance Enterography (MRE) from baseline to 12 weeks | Baseline and 12 weeks
  MRE is a non-invasive technology for measuring tissue stiffness that has been validated against liver fibrosis by biopsy; as liver stiffness by MRE increases systematically with fibrosis stage. MRE can also discriminate between patients with moderate and severe fibrosis (grades 2-4) and those with mild fibrosis (sensitivity, 86%; specificity, 85%). MRE will be performed during the same scan for adipose tissue on the research-dedicated 3.0 Tesla GE Scanner equipped with the Mayo Clinic MRE apparatus, and synchronized motion-encoded GRE sequence, based on published validation studies.
Total body fat, soft lean tissue, and bone mineral content by dual-energy x-ray absorptiometry (DXA) at baseline | Baseline
  Total body fat, soft lean tissue, and bone mineral content will be measured by dual energy x-ray absorptiometry (DXA) using a Hologic QDR 5400 densitometer (Hologic, Inc., Bedford, MA).
Total body fat, soft lean tissue, and bone mineral content by dual-energy x-ray absorptiometry (DXA) at 12 weeks | 12 weeks
  Total body fat, soft lean tissue, and bone mineral content will be measured by dual energy x-ray absorptiometry (DXA) using a Hologic QDR 5400 densitometer (Hologic, Inc., Bedford, MA).
Change in total body fat, soft lean tissue, and bone mineral content by dual-energy x-ray absorptiometry (DXA) from baseline to 12 weeks | Baseline and 12 weeks
  Total body fat, soft lean tissue, and bone mineral content will be measured by dual energy x-ray absorptiometry (DXA) using a Hologic QDR 5400 densitometer (Hologic, Inc., Bedford, MA).
Liver enzymes by fasting blood analysis at baseline | Baseline
  A fasting blood sample will be taken at the baseline visit (during the OGTT) for determination of excessively elevated liver enzymes and risk of hereditary liver disease (ALT>300 IU).
Liver enzymes by fasting blood analysis at 12 weeks | 12 weeks
  A fasting blood sample will be taken at 12 weeks (during the OGTT) for determination of excessively elevated liver enzymes and risk of hereditary liver disease (ALT>300 IU).
Change in liver enzymes by fasting blood analysis from baseline to 12 weeks | Baseline and 12 weeks
  A fasting blood sample will be taken at the baseline visit and 12 weeks (during the OGTT) for determination of excessively elevated liver enzymes and risk of hereditary liver disease (ALT>300 IU).
Fasting glucose at baseline | Baseline
  A fasting blood sample will be taken at the baseline visit (during the OGTT) for determination of elevated fasting glucose (>126 mg/dL) and risk of type 2 diabetes.
Fasting glucose from 12 weeks | 12 weeks
  A fasting blood sample will be taken at the 12 week visit (during the OGTT) for determination of elevated fasting glucose (>126 mg/dL) and risk of type 2 diabetes.
Change in fasting glucose from baseline to 12 weeks | Baseline and 12 weeks
  A fasting blood sample will be taken at the baseline and 12 week visit (during the OGTT) for determination of elevated fasting glucose (>126 mg/dL) and risk of type 2 diabetes.
Insulin and glucose response to an oral glucose challenge at baseline | Baseline
  Glucose tolerance as well as insulin secretion and clearance will be determined during a standard 2-hour oral glucose tolerance test using a glucose load of 1.75g per kg of body weight to a maximum of 75g glucose dissolved in water. Samples will be drawn at 0, 15, 30, 60, 90 and 120 minutes and will be assayed for glucose, insulin, and C-peptide.
Insulin and glucose response to an oral glucose challenge at 12 weeks | 12 weeks
  Glucose tolerance as well as insulin secretion and clearance will be determined during a standard 2-hour oral glucose tolerance test using a glucose load of 1.75g per kg of body weight to a maximum of 75g glucose dissolved in water. Samples will be drawn at 0, 15, 30, 60, 90 and 120 minutes and will be assayed for glucose, insulin, and C-peptide.
Change in insulin and glucose response to an oral glucose challenge at baseline and 12 weeks | Baseline and 12 weeks
  Glucose tolerance as well as insulin secretion and clearance will be determined during a standard 2-hour oral glucose tolerance test using a glucose load of 1.75g per kg of body weight to a maximum of 75g glucose dissolved in water. Samples will be drawn at 0, 15, 30, 60, 90 and 120 minutes and will be assayed for glucose, insulin, and C-peptide.
Lipids at baseline | Baseline
  The fasting blood sample will be assessed for lipid composition.
Lipids at 12 weeks | 12 weeks
  The fasting blood sample will be assessed for lipid composition.
Change in lipids from baseline to 12 weeks | Baseline and 12 weeks
  The fasting blood sample will be assessed for lipid composition.
Adipokines at baseline | Baseline
  The fasting blood sample will be assessed for adipocytokines.
Adipokines at 12 weeks | 12 weeks
  The fasting blood sample will be assessed for adipocytokines.
Change in adipokines from baseline to 12 weeks | Baseline and 12 weeks
  The fasting blood sample will be assessed for adipocytokines.
Inflammatory markers at baseline | Baseline
  The fasting blood sample will be assessed for inflammatory markers.
Inflammatory markers at 12 weeks | 12 weeks
  The fasting blood sample will be assessed for inflammatory markers.
Change in inflammatory markers from baseline to 12 weeks | Baseline and 12 weeks
  The fasting blood sample will be assessed for inflammatory markers.
Hormones at baseline | Baseline
  The fasting blood sample will be assessed for hormones.
Hormones 12 weeks | 12 weeks
  The fasting blood sample will be assessed for hormones.
Change in hormones from baseline to 12 weeks | Baseline and 12 weeks
  The fasting blood sample will be assessed for hormones.
Blood pressure at baseline | Baseline
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes. Three readings of blood pressure will be obtained and the average of the two last readings will be recorded.
Blood pressure at 12 weeks | 12 weeks
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes. Three readings of blood pressure will be obtained and the average of the two last readings will be recorded.
Change in blood pressure from baseline to 12 weeks | Baseline and 12 weeks
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes. Three readings of blood pressure will be obtained and the average of the two last readings will be recorded.
Resting heart rate at baseline | Baseline
  Resting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes. Three readings of heart rate will be obtained and the average of the two last readings will be recorded.
Resting heart rate at 12 weeks | 12 weeks
  Resting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes. Three readings of heart rate will be obtained and the average of the two last readings will be recorded.
Change in resting heart rate from baseline to 12 weeks | Baseline and 12 weeks
  Resting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes. Three readings of heart rate will be obtained and the average of the two last readings will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, Principal Investigator — University of Southern California; Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Diabetes & Obesity Research Institute, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt KA, Jones RB, Rios C, Corona Y, Berger PK, Plows JF, Alderete TL, Fogel J, Hampson H, Hartiala JA, Cai Z, Allayee H, Nayak KS, Sinatra FR, Harlan G, Pickering TA, Salvy SJ, Mack WJ, Kohli R, Goran MI. Clinical Intervention to Reduce Dietary Sugar Does Not Affect Liver Fat in Latino Youth, Regardless of PNPLA3 Genotype: A Randomized Controlled Trial. J Nutr. 2022 Jul 6;152(7):1655-1665. doi: 10.1093/jn/nxac046. PMID 35218194